CLINICAL TRIAL: NCT06787573
Title: Appendectomy in Elderly
Brief Title: Complications After Appendectomy in Elderly
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof of general and laparoscopic surgery, Zagazig University
Other Study IDs: appendectomy in elderly
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Appendectomy
Keywords: appendectomy;elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: postoperative complications
- Group B: No postoperative complications

SUMMARY:
this study evaluate postoperative complications after appendectomy

ELIGIBILITY:
Inclusion Criteria:

* elderly patients with AA

Exclusion Criteria:

* conservative treatment, psychological factors

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients with AA
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative complications | 30 days
  percentage of complications after surgery

SECONDARY OUTCOMES:
risk factors for complications | 30 days
  COVID-19 is a risk factor

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Habeeb TAAM, Hussain A, Bueno-Lledo J, Gimenez ME, Aiolfi A, Chiaretti M, Kryvoruchko IA, Manangi MN, Elias AA, Adam AAM, Gadallah MA, Ahmed SMA, Khyrallh A, Alsayed MH, Awad ETK, Ibrahim EA, Elshafey MH, Labib MF, Badawy MHM, Teama SRA, Seleem A, Abo Alsaad MI, Ali AK, Elbelkasi H, Abou Zaid MA, Mohamed BA, Alwadees A, El-Taher AK, Mansour MI, Yassin MA, Arafa AS, Lotfy M, Atef B, Elnemr M, Khairy MM, Abdelwanis AH, Abdelaziz AM, Mostafa A, Hamed AM, Wasefy T, Heggy IA, Nawar AMH. COVID-19-specific risk factor for early post-appendectomy complications (EPAC) in older patients: a retrospective study. Tech Coloproctol. 2025 Nov 5;29(1):188. doi: 10.1007/s10151-025-03232-1. PMID 41191115